CLINICAL TRIAL: NCT04816877
Title: Use Of Patient Controlled Analgesia For Treating The Pain Of Acute Pancreatitis: A Prospective Study
Brief Title: Use of Patient-Controlled Analgesia in Acute Pancreatitis
Acronym: PCA-AP
Status: Terminated | Type: Observational
Why Stopped: inadequate recruitment despite efforts
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Sunil Sheth, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Other Study IDs: 2021P000203
Record Dates: First submitted 2021-03-21; First posted 2021-03-25 (Actual); Results first posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-09

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Analgesics, Opioid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Patient controlled analgesia (PCA) group: Patients in this group will be allocated to the PCA arm, i.e., they will be receiving a PCA pump for administration of opioids.
  Interventions: Drug: Opioid
- Physician directed analgesia (PDA) group: Patients in this group will be allocated to the PDA arm, i.e., they will be receiving opioids administered by the nurse, as and when directed by the physician.
  Interventions: Drug: Opioid

INTERVENTIONS:
Drug: Opioid — Patients with acute pancreatitis will be divided into two groups - patient controlled analgesia (PCA) and physician-directed analgesia (PDA). Opioids are routinely administered as standard of care for treating pain associated with acute pancreatitis. Patients in the PCA group will be receiving opioids via a PCA pump, that the patient can use to self-regulate the dose and timing of drug administration. We will follow a specific protocol that has been designed by our pain physician for the PCA pump. Patients in the PDA arm will receive PRN opioids as directed by the physician, which will be administered by the nurse.

SUMMARY:
Acute pancreatitis (AP) represents a critical health concern nationwide, with estimated 274,000 admissions annually and at a cost of 2.6 billion dollars. Current treatment strategies for AP are limited to supportive care with fluid resuscitation, analgesia, nutrition and prevention of end organ damage. Abdominal pain is often the predominant symptom in patients with AP and is treated with analgesics. As there is currently no disease-specific medical treatment to change the natural history of pancreatitis, pain control remains central to the treatment of AP. Among the analgesics, opioids have been shown to be provide safe and effective pain control in patients with AP. Current literature shows that there is no difference in the risk of pancreatitis complications or clinically serious adverse events between opioids and other analgesia options. Among hospitalized AP patients, adequate pain control often requires the use of intravenous (IV) opiates in the first 24-48 hours, which can later be transitioned to oral (PO) opioids. While there are various methods of delivering opioid medications such as IV, PO, and transdermal to name a few, IV opioids are commonly administered, either on a scheduled and/or on an as needed (PRN) basis as directed by the attending physician. In contrast to the conventional, method of physician directed IV opioid delivery, patient-controlled analgesia (PCA) is a form of IV opioid medication delivery in which the patient can rapidly titrate the opioid dose to manage variable levels of pain. This modality of opioid administration is often preferred by patients and has been widely used in postsurgical and obstetric patients to effectively treat their pain. PCA allows for faster intervention on pain limiting time to treatment and peak pain levels and has also been shown to decrease total opioid dose. However, there is limited evidence in published literature assessing the feasibility of using PCA to treat the pain of AP or comparing its efficacy and safety profile compared to the more traditional physician directed analgesia. One retrospective study has shown that use of PCA was surprisingly associated with longer hospital stays and higher rates of outpatient opioid use when compared to routine physician-directed analgesia (PDA), however there are no prospective trials to study this comparison. Hence, in this study, the investigators will compare the effects of using PCA among patients with AP to that of conventional PDA.

DETAILED DESCRIPTION:
* Investigators will identify patients with AP based on the 2012 revised Atlanta criteria for diagnosis, i.e., AP is diagnosed if 2 out of the following 3 criteria are met:
* Acute onset of persistent, severe, epigastric pain often radiating to the back,
* Elevation in serum lipase or amylase to three times or greater than the upper limit of normal,
* Characteristic findings of acute pancreatitis on imaging (contrast-enhanced computed tomography [CT], magnetic resonance imaging [MRI], or transabdominal ultrasonography).
* Patients will be recruited for participation in this study while they are hospitalized with AP at Beth Israel Deaconess Medical Center. Once the patient has been transferred from the emergency department to the hospital floor, we will identify and recruit them for participation in our study.
* After obtaining informed consent from the patient, the patient will be enrolled by simple randomization to either the PCA or the PDA arm of the study. The research staff will assign patients to either the PCA arm or the PDA arm based on a standard randomization. Once, a patient has consented, the research staff will assign them to the next sequential study identidication number and corresponding study arm and let the attending hospitalist know of the result. The patient will then be enrolled in their assigned arm.
* The initial protocol for analgesic administration in each arm is as follows:

  * Recommended algorithm for physician directed analgesia (PDA) arm:

    * IV Hydromorphone 0.4 mg every 4 hours PRN for pain 4-6
    * IV hydromorphone 0.6 mg every 2 hours PRN for pain 7-10
    * Rescue IV hydromorphone 0.4 mg every 2 hours PRN for pain 4-10 = only to be given as a 'rescue dose' if patient has persistent pain despite using every 4 hours PRN IV hydromorphone (breakthrough pain)
    * Maximum opioid dosing: 1 mg per hour and 3 mg of IV hydromorphone per 4 hours
    * If patient has received more than 2 rescue doses for breakthrough pain in 12 hours or is in uncontrolled pain: Hospitalist's recommended step-up orders: IV hydromorphone 0.8 mg every 4 hours PRN 4-6
  * Recommended algorithm for patient controlled analgesia (PCA) arm:

    * IV Hydromorphone 0.1 mg every 10 minutes
    * Rescue IV hydromorphone 0.4 mg every 2 houra PRN for pain 4-6, hydromorphone 0.6 mg every 2 hours PRN for pain 7-10 = only to be given as a 'rescue' dose for if patient has persistent pain despite using PCA (breakthrough pain)
    * Maximum opioid dosing: 1 mg per hour and 3 mg of IV hydromorphone per 4 hours
    * If patient has received more than 2 rescue doses for breakthrough pain in 12 hours or is in uncontrolled pain: Hospitalist's recommended step-up orders: IV hydromorphone 0.2 mg every 10 minutes
  * Recommended for all patients:

    * PO Acetaminophen 1000 mg every 8 hours scheduled
    * IV Naloxone 40-80 mcg PRN for respiratory depression (RR<10) or significant somnolence
    * PO Benadryl 25mg every 4 hours PRN moderate to severe pruritis
  * Recommended algorithm for transition to oral:

    * PO Oxycodone 5mg every 4 hours PRN for pain 4-6
    * PO Oxycodone 10mg every 4 hours PRN for pain 7-10
    * Rescue PO Oxycodone 5mg every 2 hours PRN for pain 4-10 = only to be given as a 'rescue dose' if patient has persistent pain despite using every 4 hours PO oxycodone (breakthrough pain)
* Dosing and frequencies of medications in the above algorithms are recommendations. The recommended doses are not required for maintenance in the study and we anticipate that they may change given patient characteristics and variable response to medication, the rapidly evolving nature of acute pancreatitis, and hospitalist preferences. However, the mode of IV opioid administration (PDA vs PCA) should remain as assigned until transition to PO opioid.
* Each patient will be closely monitored for adverse events related to opioid administration to include cardiorespiratory decompensation, hemodynamic instability, nausea, vomiting, confusion, altered mental status, headache, drowsiness, etc. This monitoring will include continuous pulse oximetry in addition to vital sign measurement every 4 hours.
* The efficacy of each treatment arm to adequately control the patient's pain will be assessed with scheduled use of the Numeric Rating Scale (NRS) every 4 hours by the nursing staff. Pain rating on the NRS will be documented by the nursing staff after each assessment. In an NRS, patients are asked to circle the number between 0 and 10 that fits best to their pain intensity. Zero usually represents 'no pain at all' whereas 10 represents 'the worst pain ever possible'.
* Likert scale of 1 to 10 (1 = Very poor, 10= excellent) will be used to grade overall patient satisfaction with pain control.
* Once each patient's pain is well controlled on IV opioid administration (as determined by the attending physician) and they can tolerate intake by mouth, transition from IV to PO opioid medication can be made in each arm by the attending physician. If the patient is unable to tolerate either the PDA or the PCA arm for any reason and requires switching over to the other arm as part of his/her clinical care, they will be withdrawn from the study and their data will be excluded while analyzing the results. AP has a variable course and may require IV opioids after transition to PO opioids. The modality of IV opioid administration will revert to the assigned treatment arm.
* Other aspects of each patient's routine clinical care will continue as per the attending physician under whom the patient is admitted regardless of treatment arm status (PDA vs PCA).
* At the end of their hospital stay, investigators will document study outcomes.
* Investigators expect to enroll patients over a 36-month period from the start date of the study. Based on this, investigators expect patient enrollment to end by 4/30/2024. Investigators will plan to perform data analysis at two points: 1. Interim data analysis at a predetermined point in the study (mid-point of study), and 2. At the end of the study once patient enrollment has been completed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute pancreatitis confirmed by revised Atlanta criteria
* Admitted to the medical floor within 48 hours of emergency department arrival at Beth Israel Deaconess Medical Center (BIDMC) in Boston, Massachusetts.
* Age 18-65

Exclusion Criteria:

* Active illicit drug use
* Discharged from the emergency department
* Direct admission to ICU from emergency department
* Known allergy to opioid medications
* Age <18 or >65
* Known chronic pain syndrome or concurrent other medical condition with chronic pain
* Active encephalopathy/confusion/delirium/psychiatric illness or any other condition that limits capacity
* Known chronic opioid use
* Renal insufficiency (baseline Creatinine of >2 and/or acute kidney injury with Creatinine>3 on admission)
* Known allergy to acetaminophen or hepatic dysfunction otherwise limiting acetaminophen use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with acute pancreatitis who are admitted to our hospital (BIDMC) and meet above mentioned inclusion criteria will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2023-12-07 (Actual); Study Completion 2023-12-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were recruited from a single tertiary care center. The first patient was recruited on 2/22/2022 and the last patient on 10/17/2023.
Pre-assignment Details: All the 7 patients underwent assignment to both the treatment groups
Period: Overall Study
Arm/Group | Patient Controlled Analgesia (PCA) Group | Physician Directed Analgesia (PDA) Group
Started | 3 | 4
Completed | 2 | 4
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: We anticipated a non-parametric distribution of age which warranted description as median (IQR). Sex and ethnoracial distribution were described as frequency (percentage).
Groups:
- Total: Total of all reporting groups
Arm/Group | Physician Directed Analgesia (PDA) Group | Patient Controlled Analgesia (PCA) Group | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [54 to 67.25] | 58 [58 to 59] | 58 [56.5 to 62.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Length of Stay (Days)
Description: amount of time enrolled participants are admitted to the hospital.
Time Frame: 4-21 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Patient Controlled Analgesia (PCA) Group | Physician Directed Analgesia (PDA) Group
Number analyzed (Participants) | 3 | 4
days | 12 (4) | 9.75 (5.5)

2. Secondary Outcome: Number of Days the Patient Gets Nothing by Mouth (NPO) Before Diet is Initiated
Description: The duration of time between patient presentation and dietary advancement was noted.
Time Frame: From date of hospital admission to discharge, assessed up to 12 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Patient Controlled Analgesia (PCA) Group | Physician Directed Analgesia (PDA) Group
Number analyzed (Participants) | 3 | 4
days | 3 (0) | 6.25 (7.8)

3. Secondary Outcome: Mean Pain Scores on a Numeric Rating Scale (NRS) Over the First 24 Hours and Over Entire Course of Their Hospital Stay
Description: Mean pain scores over the first 24 hours, second 24 hours, and course of their hospital stay were recorded using a numeric rating scale which ranged from 0 to 10 where 0 is no pain and 10 is the worst pain imaginable.
Time Frame: Day 1 of hospitalization and Average Pain Score throughout entire hospital stay, assessed up to 12 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Patient Controlled Analgesia (PCA) Group | Physician Directed Analgesia (PDA) Group
Number analyzed (Participants) | 3 | 4
units on a scale
  Mean NRS over 24 hrs | 5.5 (0) | 5.6 (3.14)
  NRS over entire stay | 2.1 (0) | 7 (3.46)

4. Secondary Outcome: Total Morphine Milligram Equivalent
Description: The total opioid dose for pain control was quantified through Total morphine milligram equivalent which was calculated based on the standardized conversion of opioids.
Time Frame: Through hospital stay, an average of 5-7 days
Measure: Mean (Standard Deviation); unit: morphine milligram equivalents
Arm/Group | Patient Controlled Analgesia (PCA) Group | Physician Directed Analgesia (PDA) Group
Number analyzed (Participants) | 3 | 4
morphine milligram equivalents | 110 (0) | 291 (324.8)

5. Secondary Outcome: Time to Transition to PO Opioids
Description: The time from the transition of IV opioids to PO opioids was recorded.
Time Frame: Through hospital stay, an average of 5-7 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Patient Controlled Analgesia (PCA) Group | Physician Directed Analgesia (PDA) Group
Number analyzed (Participants) | 3 | 4
days | 2 (0) | 7.67 (8.9)

6. Secondary Outcome: Number of Participants With Opioid-related Adverse Events
Description: Opioid-related adverse events were prospectively collected.
Time Frame: Through hospital stay, an average of 5-7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Physician Directed Analgesia (PDA) Group | Patient Controlled Analgesia (PCA) Group
Number analyzed (Participants) | 4 | 3
Participants | 0 | 0

7. Secondary Outcome: Number of Participants With Use of Naloxone and Antiemetics
Description: Use of naloxone and antiemetics was noted for each recruited subject.
Time Frame: Through hospital stay, an average of 5-7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Controlled Analgesia (PCA) Group | Physician Directed Analgesia (PDA) Group
Number analyzed (Participants) | 3 | 4
Participants | 0 | 0

8. Secondary Outcome: Number of Participants With ICU Transfer
Description: Transfer of patients to the intensive care unit was prospectively noted.
Time Frame: Through hospital stay, an average of 5-7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Controlled Analgesia (PCA) Group | Physician Directed Analgesia (PDA) Group
Number analyzed (Participants) | 3 | 4
Participants | 0 | 0

9. Secondary Outcome: Number of Participants With 30-day Readmission
Description: The 30-day readmission rates were prospectively noted.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Controlled Analgesia (PCA) Group | Physician Directed Analgesia (PDA) Group
Number analyzed (Participants) | 3 | 4
Participants | 1 | 0

10. Secondary Outcome: All-cause Inpatient Mortality and Opioid-related Inpatient Mortality
Description: All-cause inpatient mortality and opioid-related inpatient mortality were recorded.
Time Frame: Through hospital stay, an average of 5-7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Controlled Analgesia (PCA) Group | Physician Directed Analgesia (PDA) Group
Number analyzed (Participants) | 3 | 4
Participants | 0 | 0

11. Secondary Outcome: 30-day Mortality
Description: 30-day mortality was prospectively noted.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Physician Directed Analgesia (PDA) Group | Patient Controlled Analgesia (PCA) Group
Number analyzed (Participants) | 4 | 3
Participants | 0 | 0

12. Secondary Outcome: Daily Morphine Milliequivalents on Discharge
Description: Daily morphine milliequivalents on discharge were recorded prospectively
Time Frame: Through hospital stay, an average of 5-7 days
Measure: Mean (Standard Deviation); unit: morphine milligram equivalents
Arm/Group | Patient Controlled Analgesia (PCA) Group | Physician Directed Analgesia (PDA) Group
Number analyzed (Participants) | 3 | 4
morphine milligram equivalents | 15 (25.8) | 11.25 (22.5)

ADVERSE EVENTS:
Time Frame: 1 months
Arm/Group | Patient Controlled Analgesia (PCA) Group | Physician Directed Analgesia (PDA) Group
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/4

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/77/NCT04816877/Prot_SAP_000.pdf